CLINICAL TRIAL: NCT03375645
Title: Montefiore Opioid and Pain Study
Acronym: MOPS
Status: Completed | Type: Observational
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-8419
Record Dates: First submitted 2017-12-12; First posted 2017-12-18 (Actual); Last update posted 2022-02-17 (Actual); Status verified 2022-02

CONDITIONS: Acute Pain
MeSH Terms: conditions — Acute Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Any oral opioid — Emergency department patients who receive a prescription for an oral opioid

SUMMARY:
This study will determine pain and opioid outcomes 3 & 6 months after an emergency department visit for acute pain. This is an observational study. Patients are enrolled during an ED visit and followed by telephone 3 & 6 months later. Opioid databases will also be reviewed.

ELIGIBILITY:
Inclusion Criteria:

* Adults seen in the emergency department for acute, new-onset pain, defined as: 1)localized pain duration < 10 days and 2) prior to the acute episode, the patient has not had this type of pain in the preceding six months
* Upon emergency department discharge, the patients is prescribed an opioid for pain

Exclusion Criteria:

* Any prescribed opioid use within the previous six months including methadone and buprenorphine

  * Frequent use of any analgesic medication (Use of any analgesic >10 days per month prior to the onset of acute pain)
  * Not available for follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Emergency department patients who are evaluated for acute pain and are prescribed an oral opioid
Sampling Method: Non-Probability Sample
Enrollment: 462 (Actual)
Dates: Start 2017-11-08 (Actual); Primary Completion 2022-02-15 (Actual); Study Completion 2022-02-15 (Actual)

PRIMARY OUTCOMES:
Subsequent opioid prescription | 6 months
  All participants in this study received an opioid prescription at the time of discharge from the emergency department. Using a review of a prescription monitoring database, this study will determine whether participants received a subsequent prescription for an opioid medication.
Chronic pain in the affected body part | 6 months
  An affirmative response to the following question: its been about 180 days since you left the ER. Have you had pain on more than 50% of these days?

SECONDARY OUTCOMES:
3 item PEG score | 3 months and 6 months after ED discharge
  This is a validated pain questionnaire with 3 questions
Pain description | 3 months and 6 months after ED discharge
  Severe, moderate, mild or no pain

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Friedman, MD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No